CLINICAL TRIAL: NCT01461265
Title: Cryoablation for the Palliation of Painful Bone Metastases
Brief Title: Safety and Efficacy of Cryoablation for the Palliation of Painful Bone Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CUC10-BNE11
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Pain; Neoplasm Metastasis
Keywords: Painful bone metastases; Bone metastases; Metastatic bone tumors; Metastatic bone pain; Cryoablation; Cryotherapy; Cryosurgery
MeSH Terms: conditions — Pain; Neoplasm Metastasis; Bone Neoplasms | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Other): All subjects will have cryoablation on one or two painful metastatic bone tumors.
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — For cryoablation in the palliation of painful bone metastases, subject preparation, anesthesia, intra-operative monitoring, and postoperative management are identical to those of standard cryoablation routinely performed at all clinical centers participating in this study and are at the discretion of the investigator.
  Other Names: Cryotherapy; Cryosurgery; Visual-ICE Cryoablation System; SeedNet Cryoablation System; PresIce Cryoablation System; IceRod Cryoablation Needle; IceRod PLUS Cryoablation Needle; IceEDGE 2.4 Cryoablation Needle; IceSeed Cryoablation Needle; IceSphere Cryoablation Needle

SUMMARY:
This study will evaluate the safety and efficacy of cryoablation therapy for relief of pain associated with metastatic bone tumors.

DETAILED DESCRIPTION:
Patients with painful bone metastases who meet the eligibility criteria and who have been determined to be an appropriate candidate for cryoablation therapy will be offered enrollment into the study. Cryoablation is the process of destroying tissue by the application of extremely cold temperatures. Galil Medical Cryoablation Systems are used as a surgical tool in the fields of general surgery, dermatology (skin), neurology (nerves), chest surgery (including lung), Ears-Nose-Throat (ENT), gynecology, oncology (cancer), proctology (colon/rectal) and urology (kidney).

Patients agreeing to participate will read and sign an informed consent form and thus become subjects in the study. Treatment will be performed using a Galil Medical cryoablation system and Galil Medical cryoablation needles. Subjects will be followed for up to 24 weeks (6 months) for palliation of pain, quality of life and analgesic usage. Baseline and follow-up data will be collected for each subject via a web-based electronic data collection tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Metastatic bone disease with metastatic disease previously confirmed by prior biopsy; or Metastatic bone disease previously confirmed on imaging [e.g. computed tomography (CT) or magnetic resonance imaging (MRI)] with known (biopsied) primary disease (primary bone cancer is excluded)
* Current analgesic therapies have failed OR the subject is experiencing intolerable side effects
* Unremitting pain that resulted in a return visit to the oncologist. The 'worst pain' in the last 24 hours must be reported to be 4 or above on a scale of 0 (no pain) to 10 (pain as bad as subject can imagine) despite pharmaceutical pain management
* Pain must be from one or two painful metastatic sites in the bone that is amenable to cryoablation with CT or MRI (additional less painful metastatic sites may be present)
* Pain from the reported one or two metastatic sites must correlate with an identifiable tumor on CT, MRI, or ultrasound (US) imaging
* Tumors must be suitable for cryoablation
* Cryoablation should be performed within 14 days of baseline evaluations
* Stable use of hormonal therapy (no changes within 4 weeks prior to the cryoablation procedure)
* Stable use of pain medications (no changes within 2 weeks prior to the cryoablation procedure)
* ECOG (Eastern Cooperative Oncology Group) scale performance status 0-3
* Life expectancy ≥ 2 months
* Platelet count >50,000/mm³ within 6 weeks screening
* INR (International Normalized Ratio) <1.5 within 6 weeks screening
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up
* If taking antiplatelet or anticoagulation medication, it must be able to be discontinued prior to the procedure for an appropriate amount of time (e.g., aspirin, ibuprofen, low molecular weight heparin preparations)
* Clinically suitable for cryoablation therapy

Exclusion Criteria:

* Leukemia, lymphoma, and myeloma
* Tumor involves a weight-bearing long bone of the lower extremity with the tumor causing > 50% loss of cortical bone
* Has undergone prior ablation treatment of the index tumor
* Prior radiation therapy of the index tumor <3 weeks prior to screening
* Index tumor causing clinical or radiographic evidence of spinal cord or cauda equina compression/effacement
* Anticipated treatment of the index tumor that would require iceball formation within 1.0 cm of the spinal cord, brain, other critical nerve structure, large abdominal vessel such as the aorta or inferior vena cava, bowel, or bladder
* Surgery at the tumor site or surgery involving the cryoablation-treated tumor (index tumor)
* Index tumor involves the skull (treatment of other painful tumors in subjects with skull tumors is not excluded)
* Patient currently with neutropenia (absolute neutrophil count <1000) within 6 weeks screening
* Uncontrolled coagulopathy or bleeding disorders
* Currently pregnant, nursing, or wishing to become pregnant during the study
* Active, uncontrolled infection
* Serious medical illness, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, cerebrovascular event within 6 months prior to study entry
* Concurrent participation in other experimental studies that could affect the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference in worst pain scores | 24 weeks post-cryoablation
  The endpoint for this study will be measured as follows: assessment of the effectiveness of cryoablation associated with palliation of pain in subjects with metastatic bone cancer by measuring the average difference of pre- and posttreatment worst pain in 24 hours from baseline to 24 hour, 1, 4, 12, and 24 week follow-up intervals as measured on the numeric 0 to 10 Brief Pain Inventory (BPI) scale.

SECONDARY OUTCOMES:
Cryoablation retreatments | 24 weeks post-cryoablation
  If the first cryoablation procedure effectively relieves pain but the relief wears off over time and the pain becomes unbearable, a second procedure may be performed. The number of repeat cryoablation treatments will be recorded.
Additional surgical treatments other than cryoablation | 24 weeks post-cryoablation
  If pain is not effectively relieved by the cryoablation, other surgical treatments may be performed. The number of these treatments will be recorded.
Reduced analgesic usage | 24 weeks post-cryoablation
  The number of subjects (percentage) who are able to reduce analgesic medications from baseline to 24 hours, 1, 4, 12, and 24 weeks after cryoablation will be recorded.
Time to maximal palliation of pain after cryoablation | 24 weeks post-cryoablation
  The difference in pain scores will be assessed from baseline to follow-up intervals after cryoablation will be analyzed. The interval indicating the most relief from pain will be compared across subjects.
Subject satisfaction with the amount palliation of pain obtained from cryoablation | 24 weeks post-cryoablation
  Subject satisfaction will be compared at baseline to follow-up intervals.
Number of adverse events | 30 days post-cryoablation
  The safety endpoint for this study is to assess the incidence and severity of intra-operative events, post operative adverse events, serious adverse events and unanticipated adverse device effects related to the cryoablation procedure.
Difference in average pain scores | 24 weeks post-cryoablation
  Difference in average pain scores from baseline to 24 hours, 1, 4, 12, and 24 weeks after cryoablation as measured on the numeric 0 to 10 BPI scale
Time to recurrence of worst pain | 24 weks post-cryoablation
  Time to recurrence of worst pain at or above baseline; worst pain score in the 24 week follow-up period as measured on the numeric 0 to 10 BPI scale

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Matteo, MD, Study Chair — Shands Medical Center, Jacksonville, FL
Locations (4):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- University of British Columbia, Vancouver, British Columbia, Canada
- University Hospital of Strasbourg, Strasbourg, France

REFERENCES:
- [Background] Callstrom MR, Atwell TD, Charboneau JW, Farrell MA, Goetz MP, Rubin J, Sloan JA, Novotny PJ, Welch TJ, Maus TP, Wong GY, Brown KJ. Painful metastases involving bone: percutaneous image-guided cryoablation--prospective trial interim analysis. Radiology. 2006 Nov;241(2):572-80. doi: 10.1148/radiol.2412051247. PMID 17057075
- [Background] Coleman RE. Management of bone metastases. Oncologist. 2000;5(6):463-70. doi: 10.1634/theoncologist.5-6-463. PMID 11110597
- [Background] Goetz MP, Callstrom MR, Charboneau JW, Farrell MA, Maus TP, Welch TJ, Wong GY, Sloan JA, Novotny PJ, Petersen IA, Beres RA, Regge D, Capanna R, Saker MB, Gronemeyer DH, Gevargez A, Ahrar K, Choti MA, de Baere TJ, Rubin J. Percutaneous image-guided radiofrequency ablation of painful metastases involving bone: a multicenter study. J Clin Oncol. 2004 Jan 15;22(2):300-6. doi: 10.1200/JCO.2004.03.097. PMID 14722039
- [Background] Callstrom MR, Charboneau JW, Goetz MP, Rubin J, Wong GY, Sloan JA, Novotny PJ, Lewis BD, Welch TJ, Farrell MA, Maus TP, Lee RA, Reading CC, Petersen IA, Pickett DD. Painful metastases involving bone: feasibility of percutaneous CT- and US-guided radio-frequency ablation. Radiology. 2002 Jul;224(1):87-97. doi: 10.1148/radiol.2241011613. PMID 12091666
- [Background] Simon CJ, Dupuy DE. Percutaneous minimally invasive therapies in the treatment of bone tumors: thermal ablation. Semin Musculoskelet Radiol. 2006 Jun;10(2):137-44. doi: 10.1055/s-2006-939031. Epub 2006 Apr 5. PMID 16598666
- [Background] Ullrick SR, Hebert JJ, Davis KW. Cryoablation in the musculoskeletal system. Curr Probl Diagn Radiol. 2008 Jan-Feb;37(1):39-48. doi: 10.1067/j.cpradiol.2007.05.001. PMID 18054665